CLINICAL TRIAL: NCT04141839
Title: Safer Bars: A Cluster-Randomized Effectiveness Evaluation of Alcohol-related Sexual Violence Prevention Through Bar Staff Bystander Training
Brief Title: Evaluation of the Safer Bars Prevention Program for Sexual Assault
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mary Koss (Other)
Collaborators: Arizona State University (Other); Arizona Department of Health Services (Other Government)
Responsible Party: Sponsor-Investigator, Mary Koss, Co-Principal Investigator, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01AA027263-01 (NIH)
Record Dates: First submitted 2019-10-22; First posted 2019-10-28 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Sexual Assault Precursor Behavior

STUDY DESIGN:
Intervention Model Description: A cluster-randomized trial design with crossover to randomize participants at the bar level into intervention and delayed intervention arms.
Who Masked: Participant
Masking Description: Participants use code numbers to submit their data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Delayed intervention: baseline and 3-month assessment prior to receiving the Safer Bars training.
  Interventions: Behavioral: Safer Bars
- Intervention (Experimental): This arm with consist of bars randomized to have the Safer Bars training on their premises attended by all their liquor serving staff with assessment directly before and after training (pre/post), and at 3 and 6 months post-training follow-up.
  Interventions: Behavioral: Safer Bars

INTERVENTIONS:
Behavioral: Safer Bars — Safer Bars, a primary perpetration prevention program based on a bystander intervention model and the theory of planned behavior. Bar staff are trained to recognize and respond to sexual aggression and its precursors among patrons.

SUMMARY:
The goal is to evaluate at three sites the implementation of the Safer Bars sexual assault prevention program.

DETAILED DESCRIPTION:
Sexual violence perpetration is robustly associated with social contexts that support high levels of alcohol consumption. Beginning in 2007, the Arizona Department of Health Services (ADHS) developed and field-tested the Safer Bars curriculum with support from the CDC Rape Prevention and Education (RPE) funding program. Safer Bars is a bystander prevention training for staff of alcohol serving establishments. This application proposes a theory-driven, quasi-experimental effectiveness evaluation based at The University of Arizona. Our approach is significant because few evaluations have measured behavioral outcomes as well as the mediators that explain the observed changes in bystander behavior, or community-level outcomes associated with such interventions. Specific Aims: the specific aims are to: (1) Test a hypothesized mediational model of individual-level behavioral outcomes based on the Theory of Planned Behavior; (2) assess the effect of the program on bar-level risk management safety policies; and (3) examine the community-level impact of the Safer Bars program on reducing the number of police dispatches in areas with high densities of alcohol-serving establishments. Methods: A cluster-randomized trial design with crossover to randomize participants at the bar level into intervention and delayed intervention arms is proposed. Assessments are at baseline, completion of training, and at three and six months post-training. The sample bars will be selected within a three-mile radius of the three major Arizona universities, all of which have a high density of alcohol-serving establishments adjacent to campus. Our analytical model will assess a hypothesized moderated mediational model based in the Theory of Planned Behavior (TPB). Outcomes of interest include: (a) the extent to which Behavioral Intent, the central construct of TPB, mediates bar staff performance of intended bystander behaviors at three-month follow-up and the extent to which this relationship is moderated by personal characteristics and bar environment; (b) the effects of the program on bar-level risk management patron safety policies; and, (c) the community-level effects as demonstrated by number of police dispatches in areas with a high density of alcohol-serving establishments at baseline and at the end of the project using GIS data. With evidence of efficacy, Safer Bars is feasible for scale-up without excessive financial burden in other states, which all receive RPE funding.

ELIGIBILITY:
Inclusion Criteria:

* Both an employee and a liquor server, security official, or owner/manager of a bar randomly selected to receive Safer Bars training immediately or after an assessment only phase of 4 months and that has not participated in the Safe Bars training in the past 12 months. Accepts healthy volunteers as defined by holding active employment. Employees may opt out of training and/or assessment.

Exclusion Criteria:

* None. No liquor servers are allowed by law to be younger than 19 years old.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 681 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Koss, PhD, Principal Investigator — University of Arizona; Kelly C Davis, MSW, PhD, Principal Investigator — Arizona State University
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified responses to survey questions will be provided to qualified investigators upon request with the time frame conditions described below. Any measures used that were developed or modified by the investigators will be provided as will the study protocol, SAP, and analytic code will be provided at any point after study completion to facilitate replication studies.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Five years after study completion, or sooner if requested by journal reviewers or colleagues for purposes of writing comments or critiques.
Access Criteria: Research institution

REFERENCES:
- [Background] Davis KC, Koss MP, Lopez EC, Roberts K. Safer Bars: A cluster-randomized effectiveness evaluation of alcohol-related sexual violence prevention through bar staff bystander training. Contemp Clin Trials. 2024 May;140:107488. doi: 10.1016/j.cct.2024.107488. Epub 2024 Mar 6. PMID 38458561
- [Result] Roberts K, Davis KC, Koss MP, Lopez EC. Feasibility and Acceptability of a Bar-Staff Bystander Intervention Training Program for Reducing Sexual Aggression. J Stud Alcohol Drugs. 2025 Mar;86(2):238-245. doi: 10.15288/jsad.24-00031. Epub 2024 Oct 15. PMID 39404150

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Staff: Delayed intervention: baseline and 3-month assessment prior to receiving the Safer Bars training.
  Safer Bars: Safer Bars, a primary perpetration prevention program based on a bystander intervention model and the theory of planned behavior. Bar staff are trained to recognize and respond to sexual aggression and its precursors among patrons.
- Intervention Staff: This arm with consist of bar staff randomized to have the Safer Bars training on their premises attended by all their liquor serving staff with assessment directly before and after training (pre/post), and at 3 and 6 months post-training follow-up.
  Safer Bars: Safer Bars, a primary perpetration prevention program based on a bystander intervention model and the theory of planned behavior. Bar staff are trained to recognize and respond to sexual aggression and its precursors among patrons.
- Control Managers: Delayed intervention: baseline and 3-month assessment prior to receiving the Safer Bars training.
  Safer Bars: Safer Bars, a primary perpetration prevention program based on a bystander intervention model and the theory of planned behavior. Bar managers are trained to recognize and change bar policies and environment to reduce sexual aggression and its precursors among patrons.
- Intervention Managers: This arm will consist of bar managers randomized to have the Safer Bars training on their premises attended by all their liquor serving staff with assessment directly before and after training (pre/post), and at 3 months post-training follow-up.
  Safer Bars: Safer Bars, a primary perpetration prevention program based on a bystander intervention model and the theory of planned behavior. Bar managers are trained to recognize and change bar policies and environment to reduce sexual aggression and its precursors among patrons.
Period: Overall Study
Arm/Group | Control Staff | Intervention Staff | Control Managers | Intervention Managers
Started | 310 | 321 | 24 | 26
Post Training Assessment | 0 (Milestone not applicable because control group did not receive training) | 259 | 0 | 24
3 Month Follow up Complete | 242 | 257 | 14 | 21
6 Month Follow up | 0 (Milestone not applicable because control group did not receive 6 month follow up) | 227 | 0 (Milestone not applicable because control managers did not receive 6 month follow up) | 0 (Milestone not applicable because intervention managers did not receive 6 month follow up)
Completed | 242 | 278 | 14 | 21
Not Completed | 68 | 43 | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Intervention Staff: This arm will consist of staff randomized to have the Safer Bars training on their premises attended by all their liquor serving staff with assessment directly before and after training (pre/post), and at 3 and 6 months post-training follow-up.
  Safer Bars: Safer Bars, a primary perpetration prevention program based on a bystander intervention model and the theory of planned behavior. Bar staff are trained to recognize and respond to sexual aggression and its precursors among patrons.
- Intervention Managers: This arm with consist of managers randomized to have the Safer Bars training on their premises attended by all their liquor serving staff with assessment directly before and after training (pre/post), and at 3 months post-training follow-up.
  Safer Bars: Safer Bars, a primary perpetration prevention program based on a bystander intervention model and the theory of planned behavior. Bar managers are trained to recognize and change bar policies and environment to reduce sexual aggression and its precursors among patrons.
- Total: Total of all reporting groups
Arm/Group | Control Staff | Intervention Staff | Control Managers | Intervention Managers | Total
Number analyzed (Participants) | 310 | 321 | 24 | 26 | 681
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 310 | 321 | 24 | 26 | 681
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Male | 154 | 179 | 17 | 13 | 363
  Sex/Gender: Female | 142 | 126 | 5 | 13 | 286
  Sex/Gender: Not reported | 14 | 16 | 2 | 0 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 160 | 144 | 15 | 16 | 335
  Multiracial | 18 | 17 | 0 | 0 | 35
  Hispanic/Latino | 98 | 106 | 6 | 8 | 218
  Black/African-American | 5 | 18 | 0 | 1 | 24
  American Indian/Alaska Native | 3 | 15 | 0 | 0 | 18
  Middle Eastern/North African | 0 | 0 | 0 | 0 | 0
  Native Hawaiian/Pacific Islander | 1 | 2 | 0 | 0 | 3
  Asian | 6 | 4 | 0 | 1 | 11
  Not reported | 19 | 15 | 3 | 0 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported Always Intervening Behavior at 6 Months
Description: Self-reported survey items measuring actual behavior (action taken) in response to observation of sexual aggression in the bar environment will be analyzed to identify significant differences post-intervention.
Time Frame: at baseline and up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Staff | Intervention Staff
Number analyzed (Participants) | 310 | 321
Participants | 207 | 239

2. Primary Outcome: Did Not Offer Promotions Aimed at Attracting Female Patrons Post-intervention
Description: Self-reported survey items completed by bar owners/managers regarding promotions aimed at attracting female patrons
Time Frame: at baseline and up to 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Control Managers: Delayed intervention: baseline and 3-month assessment prior to receiving the Safer Bars training.
  Safer Bars: Safer Bars, a primary perpetration prevention program based on a bystander intervention model and the theory of planned behavior. Bar managers are trained to recognize and change bar policies and environments to reduce sexual aggression and its precursors among patrons.
Arm/Group | Control Managers | Intervention Managers
Number analyzed (Participants) | 14 | 21
Participants | 13 | 15

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/335 | 0/346
Serious Adverse Events (participants affected / at risk) | 0/335 | 0/346
Other Adverse Events (participants affected / at risk) | 0/335 | 0/346

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT04141839/Prot_SAP_000.pdf